CLINICAL TRIAL: NCT06405555
Title: Midodrine in Heart Failure With Reduced Ejection Fraction With Hypotension: A Pilot, Open-label, Randomized Controlled Trial
Brief Title: Midodrine in Heart Failure With Reduced Ejection Fraction With Hypotension
Acronym: MIDOH-HF-P
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5784
Record Dates: First submitted 2024-04-25; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Hypotension; LV Dysfunction
Keywords: Heart Failure; GDMT; Midodrine
MeSH Terms: conditions — Hypotension; Ventricular Dysfunction, Left; Heart Failure | interventions — Midodrine

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 fashion to either the treatment arm (midodrine + standard of care) or control (no-midodrine, standard of care).
Masking Description: The study is open label and neither the study participant, research team, or members within the circle of care of the patient will be blinded to the randomization/treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Midodrine treatment (Experimental): Patients randomized to receive midodrine for up to 5 days in hospital at escalating doses starting at 2.5 mg po TID x 1 day, 5.0 mg po TID x 1 day, 7.5 mg po TID x 1 day, 10 mg po TID x 2 days. Patients may be discharged from hospital prior to completion of the full 5 day protocol. All patients in the midodrine treatment arm will receive otherwise usual standard of care treatments.
  Interventions: Drug: Midodrine Oral Tablet
- Control (No Intervention): Patients randomized to the control arm will receive usual standard of care treatments without addition of midodrine.

INTERVENTIONS:
Drug: Midodrine Oral Tablet — Exposure to up to 5 days of midodrine (or until hospital discharge) in hospital at escalating doses with the following protocol: 2.5 mg po TID x 1 day, 5.0 mg po TID x 1 day, 7.5 mg po TID x 1 day, 10 mg po TID x 2 days.
  Other Names: Midodrine hydrochloride
  Arms: Midodrine treatment

SUMMARY:
The evidence-based pharmacologic treatments available for patients with heart failure with reduced ejection fraction (HFrEF) has been established over the last few decades of cardiovascular research. These treatments, termed Foundational Guideline-Directed-Medical Therapies (GDMT), prolong patient life, improve patient-reported symptoms, and reduce hospitalizations for heart failure. A direct effect of most medication classes encompassed within GDMT is the reduction in blood pressure due to their mechanisms of action. In addition, as patients with HFrEF become more advanced in their disease, a significant proportion develop hypotension related to pump failure and autonomic dysfunction, amongst other possible mechanisms. As a result, a significant proportion of HFrEF patients are not optimized on GDMT with hypotension as their limiting barrier that would otherwise have served to improve their heart function, heart failure symptoms, and mortality. Currently, there does not exist any evidence-based strategies to address the problem of hypotension in HFrEF patients who are not optimized on GDMT.

Midodrine is an alpha-adrenergic agonist (α1-AR) that exerts its effects on peripheral venous and arteriolar vasculature to increase blood pressure. This medication has been used off-label by some clinicians in the hypotensive HFrEF population to increase blood pressure and has been reported to have beneficial effects in improving GDMT utilization as well as increasing left ventricular ejection fraction (LVEF) in published case reports/case series. There does not exist any randomized prospective data on the use of midodrine in the hypotensive HFrEF population. The investigators' objective is to complete the first open-label, randomized control trial of midodrine in the hypotensive HFrEF population to demonstrate feasibility in performing a trial in this patient population and to show efficacy in increasing blood pressure without associated harm. The results of this trial will be used as the foundation and rationale for future studies assessing the impact of midodrine use on GDMT utilization as well as hard cardiovascular outcomes in the hypotensive HFrEF population, including hospitalizations for heart failure and mortality.

DETAILED DESCRIPTION:
This will be a pilot, open-label, randomized controlled trial with the intervention/treatment being midodrine in hospitalized patients with HFrEF. The comparator/control arm will be patients following standard of care, which is to undergo no further pharmacologic intervention directed at hypotension unless clinically indicated. Patients who meet inclusion criteria will be randomized (1:1) to either midodrine group or control group, which will occur at the time of recruitment. In the treatment group, patients will receive midodrine for a total planned duration of up to 5 days, or until hospital discharge, whichever comes first. The midodrine will initially be started at 2.5 mg po TID for 1 day, followed by 5.0 mg po TID x 1 day, 7.5 mg po TID x 1 day, and 10 mg po TID x 2 days. Side effects reported by patients and any adverse drug events will be documented. At the end of the inpatient study period, continuation of midodrine off-label will be at the treating clinician's discretion in the treatment arm.

For patients discharged home less than 1 week from the exposure period, patients will be followed for 2 weeks with the Telehome monitoring program (THM), which is a virtual outpatient service intended to closely follow heart failure patients, to monitor blood pressure, heart rate, weight and adverse events or side effects. For patients discharged home between 1 to 2 weeks from the exposure period, they will be followed for 1 week with THM. For patients discharged after 2 or more weeks from the exposure period, no THM follow-up will occur. Frequency of THM follow-up, as well as inpatient monitoring parameters is as outlined in the "Data Capture" section.

Key clinical measurements will be obtained in both treatment and control arms including blood pressure measurements (every 6 hours while awake, with each measurement in the treatment arm consisting of BP measured 1 hour after the administration of midodrine dose and in the supine position. For patients in the control arm, a similar frequency of blood pressures will be obtained at pre-specified times), NT-proBNP at the time of recruitment (Day 0, prior to administration of midodrine in treatment arm) and after 5 days (ie. Sample obtained at time of last dose at Day 4 or at Day 5) or hospital discharge (whichever comes first). Safety outcomes will be monitored for and assessed. The study will be open-label and neither the patient nor the treating physicians will be blinded in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years of age.
* LVEF <= 40 % within the last 3 months as determined by any one of: Transthoracic echocardiogram, transesophageal echocardiogram, cardiac magnetic resonance imaging, MUGA scan, angiogram with left ventriculogram.
* AHA/ACC Stage B or C Heart Failure
* Hospitalized patients in the ward setting OR in the cardiac intensive care unit (who are >= 48 hours after their last dose of vasopressor or inotrope).
* Seated upright or supine SBP <= 100 mmHg on two or more consecutive BP measurements separated by at least 8 hours

Exclusion Criteria:

* Patient OR substitute decision-maker (SDM) unwilling or unable to provide informed consent
* Documented allergy or intolerance to midodrine
* Treatment for active infection (either documented infection or empiric treatment) with antimicrobials at the time of recruitment.
* Current use OR any use within the last 48 hours of an intravenous inotrope or vasopressor medication OR the need for IV inotrope or vasoproessor use to treat hypotension
* Patient within 72 hours of an acute coronary syndrome.
* Heart transplant recipient.
* Presence of temporary or durable mechanical circulatory support device.
* Severe valvular disease expected to be intervened upon during the incident hospitalization.
* Hyperkalemia >= 5.5 mmol/L.
* Baseline eGFR (as calculated by the CKD-EPI method) <= 20 mL/min/1.73 m2 as measured within the last 3 months.
* A treatable cause for hypotension, including but not limited to: hypovolemia (eg. Bleeding, overdiuresis, poor oral intake), obstructive shock, sepsis, adrenal insufficiency.
* Clinical diagnosis of ongoing cardiogenic shock, or diagnosed as defined in SHOCK trial: sBP <= 90 mmHg with evidence of end-organ hypoperfusion (cool extremities, urine output < 30 mL/hr, HR > 60 bpm, or elevated lactate >=3.5 mmol/L), invasive hemodynamic measurements (if available) of CI <= 2.2 L/min/m2 and a pulmonary capillary wedge pressure (PCWP) of >=15 mmHg.
* Pregnant patient.
* Anticipated patient discharge in less than two days from enrolment (ie. less than 6 anticipated doses of midodrine, if randomized to treatment/intervention arm).
* Acute brain pathology (including, but not limited to intracranial hemorrhage or hematoma) in which most-responsible clinician deems it unsafe to augment blood pressure.
* Untreated thyrotoxicosis
* Acute or acute on chronic liver failure
* Patient unable to take oral medications
* Bradycardia with resting heart rate less than 50 beats per minute.
* Patients on an equivalent dose of Lasix >= 80 mg IV BID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | From the date of enrolment of the first study participant, to the date of enrolment of up to 56 patients, assessed up to a maximum of 80 weeks (20 months)
  Number of participants enrolled per week
Percent enrollment | From the date of enrolment of the first study participant, to the date of enrolment of up to 56 patients, assessed up to a maximum of 80 weeks (20 months)
  Number of participants enrolled divided by number screened eligible
Randomization proportion | From the date of enrolment of the first study participant, to the date of enrolment of up to 56 patients, assessed up to a maximum of 80 weeks (20 months)
  Number of participants randomized divided by number of participants enrolled
Percentage of protocol completion | From the date of enrolment of the first study participant, to the date of enrolment of up to 56 patients, assessed up to a maximum of 80 weeks (20 months)
  Number of participants completing the study protocol divided by the number of participants randomized.
Percentage lost to follow-up | From the date of enrolment of the first study participant, to the date of enrolment of up to 56 patients, assessed up to a maximum of 80 weeks (20 months)
  Number of participants lost to follow-up divided by number of participants randomized.

SECONDARY OUTCOMES:
SBP at baseline compared to Day 4 or hospital discharge if earlier | Measures from time of enrolment (Day -1 or 0) and Day 4, or hospital discharge if earlier
  Measurement of systolic blood pressure averaged over at least two measurements per day at study enrolment compared to average systolic blood pressure averaged over at least three measures on Day 4, or hospital discharge if earlier. The measurement is numerical difference in systolic blood pressure averages (mmHg). Blood pressure measurements are both supine lying measurements.
Proportion of patients achieving sBP > 105 mmHg on Day 4 or hospital discharge if earlier | Measurement from Day 4 of study protocol, or hospital discharge if earlier
  Measurement of systolic blood pressure averaged over at least three measures on Day 4, or hospital discharge if earlier. The measurement is numerical percentage. Blood pressure measurements are both supine lying measurements.
DBP at baseline compared to Day 4 or hospital discharge if earlier | Measures from time of enrolment (Day -1 or 0) and Day 4, or hospital discharge if earlier
  Measurement of diastolic blood pressure averaged over at least two measurements per day at study enrolment compared to average diastolic blood pressure averaged over at least three measures on Day 4, or hospital discharge if earlier. The measurement is numerical difference in diastolic blood pressure averages (mmHg). Blood pressure measurements are both supine lying measurements.
NT-proBNP at baseline compared to Day 4 or hospital discharge if earlier. | Measures from time of enrolment (Day -1, or earlier if available) and Day 4, or hospital discharge if earlier
  Measurement of NT-proBNP blood test at baseline at time of study enrolment minus the measurement of NT-proBNP at Day 4 of the study protocol, or hospital discharge if earlier.
Time from randomization to hospital discharge (days). | From the date of participant randomization to the date of discharge from hospital (to home, rehabilitation or transitional institution, long-term care/nursing home), up to 4 weeks.
  Date of hospital discharge subtracted by date of study randomization, expressed in days.
Hypotension events with SBP<80 mmHg within 48 hours of discontinuation of midodrine not attributable to other reversible causes | From time of study Day 4 (or last day of midodrine exposure) up to 48 hours after last exposure.
  Blood pressure event is recorded with systolic blood pressure < 80 mmHg during the study protocol in patients on midodrine where the team involved within the participants clinical circle of care do not have other attributable reversible causes.
Number of GDMT drugs at any dosage | Days 0, 4 (or hospital discharge if earlier), and at up to 4 weeks (Day 27) at the end of the protocol..
  Average number of Guideline Directed Medical Therapy medications for HFrEF (of the following medication classes: (1) ACEi/ARB/ARNI, (2)Beta-blocker, (3) Mineralocorticoid Receptor Antagonist, (4) SGLT2i) in the midodrine group and control groups.
Number of GDMT drugs at >= 50% of goal trial dosages as outlined in clinical practice guidelines | Days 0, 4 (or hospital discharge if earlier), and at up to 4 weeks (Day 27) at the end of the protocol..
  Average number of Guideline Directed Medical Therapy medications for HFrEF (of the following medication classes: (1) ACEi/ARB/ARNI, (2)Beta-blocker, (3) Mineralocorticoid Receptor Antagonist, (4) SGLT2i) at >=50% of goal trial dosages as outlined in the CCS/CHFS 2021 HFrEF guidelines in the midodrine group and control groups.
Heart Failure Collaboratory(HFC) score | Days 0, 4 (or hospital discharge if earlier), and at up to 4 weeks (Day 27) at the end of the protocol..
  Heart Failure Collaboratory score calculated in the midodrine and control groups. Minimum 0, Maximum 8, with higher scores reflecting better outcomes.
Number of hospital re-admissions within 4 weeks of inpatient exposure period | From time of study Day 0 to 28 days (inclusive) after inpatient exposure period (up to five days).
  Number of hospital admissions in the timeframe specified in both midodrine and control groups.
Number of hospitalizations for heart failure within 4 weeks of inpatient exposure period | From time of study Day 0 to 28 days (inclusive) after inpatient exposure period (up to five days).
  Number of hospital admissions for heart failure in the timeframe specified in both midodrine and control groups.
Number of deaths within 4 weeks of protocol completion | From time of study Day 0 to 28 days (inclusive) after inpatient exposure period (up to five days).
  Number of deaths in the timeframe specified in both midodrine and control groups.
Heart rate | Physiologic parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Heart rate average measurement at baseline at time of enrolment and Day 4 (or hospital discharge if earlier) in both midodrine and control groups.
Sodium laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in mmol/L.
Potassium laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in mmol/L.
Chloride laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in mmol/L.
Bicarbonate (HCO3) laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in mmol/L.
Urea laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in mmol/L.
Creatinine laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in micromol/L (umol/L)
Alanine Transaminase (ALT) laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in U/L (Units/L)
Aspartate Transaminase (AST) laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in U/L (Units/L)
Alkaline Phosphatase (ALP) laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in U/L (Units/L)
Total Bilirubin (TBili) laboratory value | Biochemical parameters at baseline and Day 4 (if available) or hospital discharge if earlier.
  Blood test. Units in micromol/L (umol/L).

OTHER OUTCOMES:
Number of serious adverse events after initiation of midodrine. | At Day 0 (or hospital discharge if earlier) up to 48 hours after last dose of midodrine
  Defined as any untoward medical occurrence that:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity (i.e. a substantial disruption in an individual's ability to conduct normal life functions)
  * Is a congenital anomaly or birth defect
  * Other medically important condition that, based on medical judgment, may jeopardize the patient, and may require medical or surgical intervention to prevent one of the outcomes listed above
Midodrine intolerance | At Day 0 to Day 4 (or hospital discharge if earlier).
  Intolerance defined as the percentage of patients that needed to stop taking midodrine due to any AE or SAE, or other reasons as indicated by the patient.
Adverse Drug Reactions (ADR) reported after initiating midodrine | At Day 0 (or hospital discharge if earlier) up to 48 hours after last dose of midodrine
  * Supine hypertension (SBP>160 mmHg)
  * New bradycardia (if HR < 50 bpm)
  * Genitourinary symptoms (Increased urinary frequency, retention, incomplete emptying, dysuria)
  * Gastrointestinal symptoms (nausea, vomiting, abdominal pain, diarrhea)
  * Pilomotor reaction
  * Paresthesia
  * Pruritis
  * Chills
  * Worsening pain (including headache)
  * Rash
  * Other

CONTACTS AND LOCATIONS:
Overall Officials: :Lisa M Mielniczuk, MD, Principal Investigator — Ottawa Heart Institute Research Corporation

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be made available upon request to qualified researchers requesting the data for scientific analysis.